CLINICAL TRIAL: NCT03447418
Title: Multiple Breath Nitrogen Washout in Healthy Volunteers
Acronym: HV-LCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0064
Record Dates: First submitted 2018-02-19; First posted 2018-02-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Lung Clearance Index; Breath Nitrogen Washout; Healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- no treatment, open label (Other)
  Interventions: Procedure: Multiple breath nitrogen washout

INTERVENTIONS:
Procedure: Multiple breath nitrogen washout — Lung Clearance Index (LCI) will be performed in healthy volunteers with a multiple breath nitrogen washout device.

SUMMARY:
This study is designed to establish reference values of multiple breath nitrogen washout indexes in an healthy population of volunteers (from childhood to adulthood)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by participant, parent, or legal guardian
* Healthy subjects with a social insurance

Exclusion Criteria:

* History of a lung chronic disease
* Premature birth (<37th weeks of amenorrhea)
* Acute lower respiratory viral infection within 3 weeks before Multiple Breath washout

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2018-07-06 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Lung Clearance Index 2.5% (LCI 2.5%) Value | hour 1
  Multiple breath washout is a pulmonary function test that does not require patients' cooperation. It studies the number of lung volumes (turn-over) to clear a gaz such as nitrogen form the lungs. LCI 2,5 is most frequently reported outcome measure. It corresponds to the sum of the total expired lung volumes needed to decrease the initial gaz concretion to its 1/40th, divided by functional residual capacity.
  LCI can be measured in infant, preschoolers and thereafter. In order to obtain reproducible tests, three acceptable maneuvers are needed.

SECONDARY OUTCOMES:
Lung Clearance Index 5% (LCI 5%) Value | hour 1
Moment ratio M1/M0 Value | up to 1 hour
Moment ratio M0/M2 Value | up to 1 hour
Sacin value | hour 1
  assessment of distal areas function
Scond value | hour 1
  assessment of conductive areas function

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided